CLINICAL TRIAL: NCT06409013
Title: Sarcoma Resection Guided by Intraoperative Indocyanine Green Dye Fluorescence Angiography
Brief Title: Evaluation of Tumor Resection Guided by Intraoperative Indocyanine Green Dye Fluorescence Angiography in Patients With Sarcoma
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-003589; NCI-2024-03482 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-003589 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Bone Sarcoma; Soft Tissue Sarcoma
MeSH Terms: conditions — Bone Neoplasms; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients receive ICG infusion prior to undergoing scheduled resection and have medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the effectiveness of intraoperative indocyanine green dye and fluoroscopic technology in confirming negative margins after tumor removal.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the use of indocyanine green (ICG) as an intraoperative guide during bone and soft tissue sarcoma resection.

OUTLINE: This is an observational study.

Patients receive ICG infusion prior to undergoing scheduled resection and have medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven bone or soft tissue sarcoma undergoing resection

Exclusion Criteria:

* * Age less than 18

  * Chronic kidney disease
  * Anaphylaxis to dyes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy-proven bone or soft tissue sarcoma undergoing resection recruited through Mayo Clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of intraoperative ICG fluorescence compared to final pathology results | Baseline
  Intraoperative ICG fluorescence and deduced margins will be analyzed and compared the accuracy to final pathology margins. Negative predictive value will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T. Houdek, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials